CLINICAL TRIAL: NCT04565912
Title: Efficacy of Sage Extract or Chlorohexidine Mouthwashes on Streptococcus Mutans Pathogenicity by Real-time Polymerase Chain Reaction (PCR) in High Caries Risk Patients : A Randomized Clinical Trial
Brief Title: Streptococcus Mutans Pathogenicity by Real-time Polymerase Chain Reaction (PCR) in High Caries Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Fayez Shebl Diab, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20788
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-09

CONDITIONS: Streptococcus Mutans

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sage extract mouthwash (Experimental): Natural product mouthwash
  Interventions: Drug: Sage extract mouthwash
- Chlorohexidine mouthwash (Active Comparator): Synthetic mouthwash
  Interventions: Drug: Chlorohexidine based mouthwash

INTERVENTIONS:
Drug: Sage extract mouthwash — Patients will be exposed to sage extract mouthwash and will be instructed to use 10 ml of sage extract mouthwash 2 times per day for 1 minute, such a regimen will be continued for one month.
  Other Names: Natural product mouthwash
  Arms: Sage extract mouthwash
Drug: Chlorohexidine based mouthwash — Patients will be exposed to Chlorohexidine based mouthwash , and will be instructed to use 10 ml of 0.12% chlorohexidine based mouthwash 2 times per day for 1 minute, such a regimen will be continued for one month
  Other Names: Synthetic mouthwash
  Arms: Chlorohexidine mouthwash

SUMMARY:
In patients with high caries risk, will the use of sage extract or chlorohexidine based mouthwashes have an effect on the percentage recovery of Streptococcus Mutans (SM) and its pathogenicity detected by Real-Time Polymerase Chain Reaction (PCR) over one month follow up

DETAILED DESCRIPTION:
The clinical study will be held in the clinic of conservative department, Faculty of Dentistry, Cairo University. The operator in charge will be Dina Fayez Diab. Patients will be examined and selected according to inclusion and exclusion criteria, the purpose and method of the study will be explained to the selected patients for participation in the study. In the first visit , ADA caries risk assessment model will be done. Participants will be divided in to two groups according to the tested mouthwashes.

All patients will be instructed not to have a breakfast and to refrain any oral hygiene measures on the day of sample collection to avoid the influence of food consumption and contamination on the composition of saliva. The patient will sit in an erect position on the dental chair and will be given paraffin block to chew. The stimulated saliva will be collected after 2 minutes of paraffin chewing in sterile container held near the mouth. The containers will be properly labelled.

This study will be carried over one month , the saliva samples for each patients will be collected on the first dental visit. These samples will be sent to the laboratory for microbiological assessment. Patients will be provided with mouthwashes according to the tested groups and will be instructed to use it 2 times per day for 1 minute each time and no eating or drinking allowed for at least 30 minutes post rinsing. Each patient will be given the same instructions with respect to oral hygiene measures. They will be advised to continue on the same diet and will be instructed not to change their dietary habits.

Patients will come after 2 weeks for salivary samples collection and samples will be sent to laboratory for microbiological assessment. After completing the treatment for another 2 weeks , patients will come for the last dental visit to collect salivary samples which will be sent to laboratory for microbiological assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients will be recruited in this study, all volunteers participated will be medically free Age range 20-50
* Patients with high caries risk assessment according to ADA caries risk assessment model High plaque index (>score 2 )
* Non smoking patients
* Patients with normal salivary rate ( 0.3-0.4 ml/min)
* Not under antibiotic therapy either time of the study or up to the last month before the begging of the study
* Male or female patients.

Exclusion Criteria:

* patients with a compromised medical history.
* Patients with low caries risk assessment according to ADA caries risk assessment model.
* Patients with sever or active periodontal disease.
* Patients with a history of allergy to any of drugs or chemicals used in this study.
* Smoking patients
* Patients with abnormal salivary rate
* Pregnant female patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-07-06 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Total bacterial count | 1 month
  Quantitative plating ( standard plate count or SPC) will be used to determine the number of bacteria in a culture sample. SPC reveals information on viable organisms only, bacteria colonies that are seen in the plates after incubation represent only the living organisms, not dead ones

SECONDARY OUTCOMES:
Bacterial identification | 1 month
  Total extraction of DNA: Total plasmid DNA will be prepared. The solution will be centrifuged and then left at room temperature for few minutes for the phase separation. The aqueous phase containing DNA will be transferred to clean eppendorf Real-Time Polymerase Chain Reaction: the PCR will be done in 20 ul reaction volume containing : DNA template, enzymes primer and nuclease- free water. The tubes containing the PCR mixture will be transferred to the cycler apparatus. The PCR products will be analyzed in agarose gel by electrophoresis, photographed and analyzed
Total protein profile | 1 month
  Proteins can be separated according to their molecular weight by Sodium dodecyl sulphate poly acrylamide gel electrophoresis (SDS-PAGE)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Expecting to have all the data by October 2022